CLINICAL TRIAL: NCT00825396
Title: A Pilot, Open-Label, Controlled Clinical Trial of C-KAD Ophthalmic Solution in Reducing Intraocular Pressure in Patients With Ocular Hypertension
Brief Title: An Open-Label Study of an Ophthalmic Solution to Reduce Intraocular Pressure in Patients With Ocular Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chakshu Research, Inc. (Industry)
Responsible Party: Ellen Hoogeveen /Associate Director, Clinical & Regulatory Affairs, Chakshu Research, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCK-0106
Record Dates: First submitted 2009-01-16; First posted 2009-01-21 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- C-KAD Ophthalmic Solution (Experimental)
  Interventions: Drug: C-KAD Ophthalmic Solution

INTERVENTIONS:
Drug: C-KAD Ophthalmic Solution — 4 drops applied daily for 150 days

SUMMARY:
The purpose of this study is to determine the safety and tolerability of topical C-KAD Ophthalmic Solution in reducing intraocular pressure in patients with ocular hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Both eyes having intraocular pressure in the range of 22-30 mmHg at baseline
* Both eyes having best corrected visual acuity better than 20/50

Exclusion Criteria:

* Advanced glaucoma
* Closed or barely open anterior chamber or history of angle closure

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Mean change in intraocular pressure from baseline | 150 Days

CONTACTS AND LOCATIONS:
Overall Officials: Ira Wong, MD, Study Director — Chakshu Research, Inc.
Locations (1):
- Charlotte Eye, Ear, Nose & Throat Associates, Charlotte, North Carolina, United States